CLINICAL TRIAL: NCT07204782
Title: Elevated Cardiovascular Risk Scores With Diabetes Mellitus Type 2 and Their Association With Non-Invasive Visceral Adiposity Indices
Brief Title: Cardiovascular Disease CVD Constitutes a Significant Health Challenge for Individuals With Type 2 Diabetes Mellitus T2DM, Affecting Approximately 32% of This Population and Contributing Significantly to Global Mortality.Visceral Adipose Tissue VAT Accumulation Has Been Recognize
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya Ahmed Mohamed Morsy, Resident doctor, Assiut University
Other Study IDs: Visceral adiposity indices
Record Dates: First submitted 2025-09-20; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Diabete Mellitus
Keywords: cardiovascular risk scores; visceral adiposity indices; diabetes mellitus; VAT; LAP
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
calculate cardiovascular risk scores in type 2 DM patients, then estimate its association with new visceral adipose tissue indices

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) constitutes a significant health challenge for individuals with type 2 diabetes mellitus (T2DM), affecting approximately 32% of this population and contributing significantly to global mortality.Visceral adipose tissue (VAT) accumulation has been recognized as a major contributor to adverse cardiac remodelling. Unlike subcutaneous adipose tissue (SAT), VAT is metabolically active, promoting a pro-inflammatory, lipotoxic, and insulin-resistant environment that accelerates myocardial fibrosis, hypertrophy, and diastolic dysfunction. Despite its clinical significance, VAT is challenging to measure in routine practice. Advanced imaging modalities such as magnetic resonance imaging provide direct VAT assessment but it's costly, time-consuming, and impractical for large-scale screening. In contrast, traditional anthropometric measures like body mass index (BMI), waist circumference (WC), and waist-to-hip ratio (WHR) do not distinguish VAT from SAT and fail to capture the true cardiometabolic burden of visceral fat .To address these limitations, researchers have focused on developing non-invasive visceral obesity indices that combine anthropometric and laboratory-based parameters. These indices are particularly relevant for T2DM patients, as insulin resistance often occurs when fat accumulates in intra-abdominal depots and is associated with a constellation of CVD risk factors, in what is known as the metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥40 years old attending the out patients clinics
* Patients diagnosed with type 2 diabetes mellitus

Exclusion Criteria:

* Patient with a history of cardiovascular events
* Patient with type 1 diabetes or gestational diabetes.
* Pregnant women.
* Hypothyroidism,
* Cushing disease
* polycystic ovarian syndrome.
* Congestive heart failure
* chronic liver disease

  .- chronic kidney disease,
* cancer
* Current use of steroids, birth control pills, antipsychotics, antidepressants, epilepsy drugs.
* Patients with physical deformities or conditions affecting anthropometric measurements.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic patients attending Assiut university
Sampling Method: Probability Sample
Enrollment: 238 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
The prevalence of elevated 10-year cardiovascular risk scores among patients with type 2 diabetes mellitus. | 1 YEAR
  Measurement tool: WHO cardiovascular risk chart
  Unit of measure: % of patients with ≥10% predicted 10-year cardiovascular risk

SECONDARY OUTCOMES:
The correlation between cardiovascular risk scores and non-invasive visceral adiposity indices (such as LAP and VAI). | 1 YEAR
  Tools: WHO cardiovascular risk chart, LAP & VAI indices
  Unit: Correlation coefficient

OTHER OUTCOMES:
The relationship between cardiovascular risk and clinical/lifestyle factors (e.g., duration of diabetes, BMI, physical activity, smoking, blood pressure, lipid profile). | 1 YEAR
  Tools: WHO cardiovascular risk chart, clinical records, questionnaires, lab tests
  Unit: Regression / correlation coefficients

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tawfik MY, Mohamed SF, Elotla SF. Association of novel visceral obesity indices with 10-year risk of major cardiovascular events in patients with type 2 diabetes mellitus. J Egypt Public Health Assoc. 2025 May 30;100(1):12. doi: 10.1186/s42506-025-00188-w. PMID 40445502
- [Background] Wang L, Liu S, Ke J, Cao B, Wang D, Zhao Q, Gong H, Fang Y, Zheng Z, Yu C, Wu N, Ma Y, Yu K, Yang L, Zhao D. Association between metabolic visceral fat score and left ventricular hypertrophy in individuals with type 2 diabetes. Diabetol Metab Syndr. 2025 Mar 6;17(1):81. doi: 10.1186/s13098-025-01648-1. PMID 40050939
- [Background] Einarson TR, Acs A, Ludwig C, Panton UH. Prevalence of cardiovascular disease in type 2 diabetes: a systematic literature review of scientific evidence from across the world in 2007-2017. Cardiovasc Diabetol. 2018 Jun 8;17(1):83. doi: 10.1186/s12933-018-0728-6. PMID 29884191